CLINICAL TRIAL: NCT00004074
Title: A Phase I Trial of Herceptin and Interleukin-12
Brief Title: Interleukin-12 and Trastuzumab in Treating Patients With Cancer That Has High Levels of HER2/Neu
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01398; 99H0185; U01CA076576 (NIH); CDR0000067282 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-12-10; First posted 2003-10-29 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Advanced Adult Primary Liver Cancer; Anaplastic Thyroid Cancer; Bone Metastases; Carcinoma of the Appendix; Distal Urethral Cancer; Fallopian Tube Cancer; Gastrinoma; Glucagonoma; Inflammatory Breast Cancer; Insulinoma; Liver Metastases; Localized Unresectable Adult Primary Liver Cancer; Lung Metastases; Male Breast Cancer; Malignant Pericardial Effusion; Malignant Pleural Effusion; Metastatic Gastrointestinal Carcinoid Tumor; Metastatic Parathyroid Cancer; Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Newly Diagnosed Carcinoma of Unknown Primary; Occult Non-small Cell Lung Cancer; Pancreatic Polypeptide Tumor; Primary Peritoneal Cavity Cancer; Proximal Urethral Cancer; Pulmonary Carcinoid Tumor; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Adrenocortical Carcinoma; Recurrent Adult Primary Liver Cancer; Recurrent Anal Cancer; Recurrent Bladder Cancer; Recurrent Breast Cancer; Recurrent Carcinoma of Unknown Primary; Recurrent Cervical Cancer; Recurrent Colon Cancer; Recurrent Endometrial Carcinoma; Recurrent Esophageal Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Recurrent Gastric Cancer; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Islet Cell Carcinoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Pancreatic Cancer; Recurrent Parathyroid Cancer; Recurrent Prostate Cancer; Recurrent Rectal Cancer; Recurrent Renal Cell Cancer; Recurrent Salivary Gland Cancer; Recurrent Small Intestine Cancer; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Thyroid Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Recurrent Vaginal Cancer; Recurrent Vulvar Cancer; Skin Metastases; Small Intestine Adenocarcinoma; Somatostatinoma; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Adrenocortical Carcinoma; Stage III Bladder Cancer; Stage III Cervical Cancer; Stage III Colon Cancer; Stage III Endometrial Carcinoma; Stage III Esophageal Cancer; Stage III Follicular Thyroid Cancer; Stage III Gastric Cancer; Stage III Malignant Testicular Germ Cell Tumor; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Ovarian Epithelial Cancer; Stage III Pancreatic Cancer; Stage III Papillary Thyroid Cancer; Stage III Prostate Cancer; Stage III Rectal Cancer; Stage III Renal Cell Cancer; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Vaginal Cancer; Stage III Vulvar Cancer; Stage IIIA Anal Cancer; Stage IIIA Breast Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Anal Cancer; Stage IIIB Breast Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Adrenocortical Carcinoma; Stage IV Anal Cancer; Stage IV Bladder Cancer; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Endometrial Carcinoma; Stage IV Esophageal Cancer; Stage IV Follicular Thyroid Cancer; Stage IV Gastric Cancer; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Pancreatic Cancer; Stage IV Papillary Thyroid Cancer; Stage IV Prostate Cancer; Stage IV Rectal Cancer; Stage IV Renal Cell Cancer; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IVA Cervical Cancer; Stage IVA Vaginal Cancer; Stage IVB Cervical Cancer; Stage IVB Vaginal Cancer; Stage IVB Vulvar Cancer; Thyroid Gland Medullary Carcinoma; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer; Urethral Cancer Associated With Invasive Bladder Cancer; WDHA Syndrome
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Appendiceal Neoplasms; Fallopian Tube Neoplasms; Gastrinoma; Glucagonoma; Inflammatory Breast Neoplasms; Insulinoma; Breast Neoplasms, Male; Pleural Effusion, Malignant; Parathyroid Neoplasms; Adrenocortical Carcinoma; Carcinoma, Hepatocellular; Anus Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Neoplasms, Unknown Primary; Uterine Cervical Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Carcinoma, Islet Cell; Testicular Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Prostatic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Thyroid Neoplasms; Urethral Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Somatostatinoma; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Carcinoma, Medullary; Vipoma | interventions — Interleukin-12 Subunit p35; Interleukin-12; Trastuzumab

ARMS (1):
- Treatment (IL12 and trastuzumab) (Experimental): Patients receive an initial loading dose of trastuzumab IV over 90 minutes on day 1 of the first week and a maintenance dose of trastuzumab IV over 30-90 minutes on day 1 of each subsequent week. Patients receive IL-12 IV on days 2 and 5 beginning on week 3. Treatment with maintenance trastuzumab and IL-12 repeats weekly for 14 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease continue treatment for up to 38 additional weeks.
  Interventions: Biological: recombinant interleukin-12; Biological: ABI-007/carboplatin/trastuzumab

INTERVENTIONS:
Biological: recombinant interleukin-12 — Given IV
  Other Names: cytotoxic lymphocyte maturation factor; IL-12; interleukin-12; natural killer cell stimulatory factor; Ro 24-7472
Biological: ABI-007/carboplatin/trastuzumab — Given IV

SUMMARY:
Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Phase I trial to study the effectiveness of interleukin-12 and trastuzumab in treating patients who have cancer that has high levels of HER2/neu and has not responded to previous therapy

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of interleukin-12 (IL-12) when combined with trastuzumab in patients with HER2-Neu overexpressing malignancies.

II. Determine the safety of this regimen in these patients.

III. Analyze any expression of interferon-inducible genes in tumor tissues of these patients after receiving this regimen.

IV. Characterize natural killer cytokine production in patients treated with this regimen.

V. Determine serum interferon gamma levels in patients treated with this regimen.

OUTLINE:

This is a dose escalation study of interleukin-12 (IL-12).

Patients receive an initial loading dose of trastuzumab IV over 90 minutes on day 1 of the first week and a maintenance dose of trastuzumab IV over 30-90 minutes on day 1 of each subsequent week. Patients receive IL-12 IV on days 2 and 5 beginning on week 3. Treatment with maintenance trastuzumab and IL-12 repeats weekly for 14 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease continue treatment for up to 38 additional weeks.

Cohorts of 3-6 patients receive escalating doses of IL-12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

Patients are followed every 3 months for 1 year and then every 6 months thereafter for survival.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically proven Her2 overexpressing malignancy as determined by any standardized assay currently in clinical use
* Patients must have measurable or evaluable disease
* The patient must have failed standard curative and/or palliative therapies for their disease
* Life expectancy of at least 6 months
* No concurrent malignancy other than non-melanoma skin carcinoma
* Adequate hematopoietic, cardiac, renal, and hepatic function
* Calculated creatinine clearance will be used to assess renal function
* Karnofsky Performance Status index >= 70%
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; a woman of childbearing potential is defined as a female who is biologically capable of becoming pregnant
* Normal cardiac ejection fraction by echocardiogram or MUGA (i.e., greater than OSU lower limit of normal)
* Written signed informed consent; the patient must be aware that his/her disease is neoplastic in nature and willingly consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts

Exclusion Criteria:

* History of significant peripheral neuropathy or significant central nervous system disease
* Brain or central nervous system metastasis at entry
* Active or unstable cardiovascular disease or cardiac disease requiring drug or device intervention; history of coronary artery disease or congestive heart failure
* Pregnant or nursing women
* Surgery, radiotherapy, chemotherapy, or hormonal therapy during the three weeks prior to the initiation of therapy
* Exposure to any investigational drug within three weeks prior to the start of dosing
* Concurrent use of systemic corticosteroids
* Known seropositive for hepatitis B surface antigen
* Known seropositive for HIV antibody
* Serious concurrent infection requiring intravenous antibiotic therapy
* Clinically significant autoimmune disease (e.g., rheumatoid arthritis)
* Clinically significant gastrointestinal bleeding or uncontrolled peptic ulcer disease
* History of inflammatory bowel disease
* Any other major illness which, in the investigator's judgment, will substantially increase the risk associated with the patient's participation in this study
* Prior therapy with Herceptin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1999-08; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events version 2.0 (CTCAE v2.0) | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States